CLINICAL TRIAL: NCT07156500
Title: A Multicenter, Randomized, Double-Blind, Placebo- Parallel Controlled, Phase III Study to Evaluate the Efficacy and Safety of HS-20094 Injection in Subjects With Type 2 Diabetes, Inadequately Controlled With Diet and Exercise Alone
Brief Title: A Phase 3 Study of HS-20094 in Patients With T2DM Inadequately Controlled With Diet and Exercise Alone
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-20094-302
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental)
  Interventions: Drug: HS-20094 Injection
- Group B (Placebo Comparator)
  Interventions: Drug: HS-20094 Placebo Injection
- Group C (Experimental)
  Interventions: Drug: HS-20094 Injection
- Group D (Placebo Comparator)
  Interventions: Drug: HS-20094 Placebo Injection

INTERVENTIONS:
Drug: HS-20094 Injection — HS-20094 injected subcutaneously once weekly
  Arms: Group A
Drug: HS-20094 Placebo Injection — HS-20094 Placebo injected subcutaneously once weekly
  Arms: Group B
Drug: HS-20094 Injection — HS-20094 injected subcutaneously once weekly
  Arms: Group C
Drug: HS-20094 Placebo Injection — HS-20094 Placebo injected subcutaneously once weekly
  Arms: Group D

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase III clinical study to evaluate the efficacy and safety of HS-20094 injection in subjects with type 2 diabetes who have inadequate glycemic control with diet and exercise alone. The primary objective of this study is to evaluate the effectiveness of HS-20094 compared to placebo in controlling blood glucose levels after 44 weeks and 52 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, Age ≥18 years at the time of signing informed consent.
2. Diagnosed with type 2 diabetes mellitus (T2DM) for at least 90 days prior to day of screening.
3. Treatment with Diet and Exercise alone at least 90 days prior to day of screening.
4. 7.5% ≤ HbA1c ≤10.5% at screening.

Exclusion Criteria:

1. Uncontrollable hypertension(with or without antihypertensive treatment) : systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg at screening.
2. Diagnosed or suspected with type 1 diabetes mellitus, special types of diabetes or secondary diabetes.
3. History of significant hematological disorders (e.g., sickle cell disease, hemolytic anemia, myelodysplastic syndrome, etc.) or other conditions causing hemolysis or instability of red blood cells (e.g., malaria, hypersplenism, etc.).
4. Presence of an endocrine disorder or history that may significantly affect bady weight(e.g., Cushing's syndrome, hypothyroidism or hyperthyroidism, except hypothyroidism if thyroid hormone replacement dose has been stable for at least 6 months) ；
5. Severe infection, severe trauma, or moderate-to-major surgery within 4 weeks before screening.
6. Participated in clinical trials of any drug or medical device within 12 weeks prior to screening, and participation in clinical trials is defined as signing informed consent and using investigational drugs (including placebo) or investigational medical devices; Or is still in the trial drug within 5 half-lives (whichever is Longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Week 0 to Week 44
  Change from baseline in HbA1c after 44 weeks of treatment

SECONDARY OUTCOMES:
Proportion of subjects with HbA1c<7.0% and ≤6.5% | Week 0 to Week 44
  Proportion of subjects with HbA1c<7.0% and ≤6.5% after 44 weeks of treatment
Change in FPG | Week 0 to Week 44
  Change from baseline in FPG after 44 weeks of treatment
Change in body weight | Week 0 to Week 44
  Change from baseline in Change in body weight after 44 weeks of treatment
Proportion of subjects with weight loss ≥5% and ≥10% | Week 0 to Week 44
  Proportion of subjects with weight loss ≥5% and ≥10% after 44 weeks of treatment
Change in HbA1c | Week 0 to Week 52
  Change from baseline in HbA1c after 52 weeks of treatment
Proportion of subjects with HbA1c<7.0% and ≤6.5% | Week 0 to Week 52
  Proportion of subjects with HbA1c<7.0% and ≤6.5% after 52 weeks of treatment
Change in FPG | Week 0 to Week 52
  Change from baseline in FPG after 52 weeks of treatment
Change in body weight | Week 0 to Week 52
  Change from baseline in Change in body weight after 52 weeks of treatment
Proportion of subjects with weight loss ≥5% and ≥10% | Week 0 to Week 52
  Proportion of subjects with weight loss ≥5% and ≥10% after 52 weeks of treatment
Incidence and severity of adverse events | Week 0 to Week 52+4 weeks follow-up
  Severity (mild, moderate and severe) is assessed by investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China